CLINICAL TRIAL: NCT01360879
Title: Assessment of Liver FIBROsis by Real-time Tissue ELASTography in Chronic Liver Disease
Acronym: FIBROELAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kindai University (Other)
Responsible Party: Japan Liver Oncology Group, Department of Gastroenterology and Hepatology, Kinki University Faculty of Medicine
Other Study IDs: JLOG1002
Record Dates: First submitted 2011-05-21; First posted 2011-05-26 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Hepatitis B; Chronic Hepatitis C
Keywords: Hepatitis B virus; Hepatitis C virus; Chronic hepatitis; Liver cirrhosis; Liver stiffness; Liver fibrosis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis C, Chronic; Hepatitis B; Hepatitis C; Hepatitis, Chronic; Liver Cirrhosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum, liver tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a multi-center cross-sectional study in which the Real-time Tissue Elastography® measurements will be collected prospectively from patients with chronic hepatitis B or C virus presenting for liver biopsy.

DETAILED DESCRIPTION:
The aim of this study is to validate the diagnostic value of Real-time Tissue Elastography® by comparison with liver histology, serum marker or FibroScan® in chronic hepatitis B or C patients.Real-time Tissue Elastography®, biopsy and serum maker are performed.

If in the hospital they can perform FibroScan®, FobroScan® also be performed. The subjects must be scheduled for liver biopsy either prior to treatment (treatment naïve) or, if previously treated, they must have been off treatment for at least six months. The time between the Real-time Tissue Elastography® , biopsy, blood sampling and FiroScan® must not exceed four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and at least 20 years of age
* Chronic hepatitis B or Chronic hepatitis C
* Subject is willing to fast for 8 hours prior to each study visit

Exclusion Criteria:

* History of alcohol abuse (alcohol intake > 20g/day)
* Evidence or history of chronic hepatitis not caused by HBV or HCV
* During 6 months before registration to this trial has completed, nucleic acid analogue preparations or interferon therapy was performed.
* Pregnant or lactating patients
* Contraindications of liver biopsy or liver resection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic hepatitis B or C, undergoing a liver biopsy as the standard of care for their disease, will be eligible for the study. Subjects with other infectious viral diseases or chronic liver disease are excluded for study enrollment.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Correlative evaluation with liver fibrosis by Real-time Tissue Elastography® and histological diagnosis | one year
  To evaluate the correlation between Real-time Tissue Elastography® index and histological diagnosis (the gold standard for liver fibrosis), we calculate sensitivity and specificity, ROC curves.
  Sensitivity, specificity and ROC curves obtained under below stiations:
  1. liver fibrosis index diagnose of histological diagnosis F4
  2. liver fibrosis index diagnose of histological diagnosis F3 or greater
  3. liver fibrosis index diagnose of histological diagnosis F2 or greater

SECONDARY OUTCOMES:
Correlative evaluation with liver fibrosis by Real-time Tissue Elastography® and serum maker | one year
  To evaluate the correlation between Real-time Tissue Elastography® index and serum markers of hepatic fibrosis, we estimate Pearson correlation coefficient of each request.
Correlative evaluation with liver fibrosis by Real-time Tissue Elastography® and FibroScan® | one year
  To evaluate the correlation between Real-time Tissue Elastography® index and FibroScan® index, we estimate Pearson correlation coefficient of each request.

CONTACTS AND LOCATIONS:
Overall Officials: Masatoshi Kudo, Professor, Study Chair — Kinki University Faculty of Medicine
Locations (1):
- Kinki University Faculty of Medicine, Ōsaka-sayama, Osaka, Japan